CLINICAL TRIAL: NCT00897520
Title: PILOT-high Throughput-protein Profiling Analysis of Sera Collected From E1694 Patients Undergoing HDI (Arm B)
Brief Title: Biomarkers in Patients With High-Risk Melanoma Receiving High-Dose Interferon Therapy
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000585297; ECOG-E1694T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha; Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Biological: recombinant interferon alfa
Genetic: proteomic profiling
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors identify biomarkers related to cancer and predict how patients will respond to treatment.

PURPOSE: This research study is looking at biomarkers in patients with high-risk melanoma receiving high-dose interferon therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To screen serum specimens using a high throughput protein profiling platform that tests for the highest number of known biomarkers (detectable by antibodies) that could be predictors of response to interferon treatment, autoimmunity, and disease outcome in patients with high-risk melanoma undergoing high-dose interferon (IFNa2b) therapy .
* To compare soluble factors across all patients at each time point (baseline and during therapy).
* To compare pre-therapy vs post-therapy serum samples from these patients.
* To assess the kinetics of soluble factors' appearance, persistence, and disappearance during the 12 months of therapy.
* To assess whether the amount of specific soluble factors in the pre-therapy sample is predictive of response independent of therapy.
* To correlate statistically significant factors with S100 and autoimmunity in these patients.
* To confirm the data obtained with the Luminex technology.

OUTLINE: Patients are stratified according to survival (< 2 years vs > 5 years).

Blood samples collected from patients enrolled in E-1694 are analyzed using high throughput protein profiling by ELISA to compare changes in levels of putative biomarkers of interferon alfa-2b, including cytokines and paired receptors, chemokines, cell adhesion molecules, metalloproteinases, angiogenic markers, growth factors, soluble receptors, signal transduction molecules, hormones, and other biomarkers of disease and dysregulated immune processes, at baseline and during therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-risk melanoma
* Receiving interferon alfa-2b therapy in arm II of clinical trial E-1694

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E1694
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-01-14 (Actual); Primary Completion 2010-01-24 (Actual); Study Completion 2010-01-24 (Actual)

PRIMARY OUTCOMES:
Serum sample screening via high throughput protein profiling in patients undergoing therapy | 1 month
Comparison of soluble factors | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Monica Panelli, PhD, Study Chair — University of Pittsburgh